CLINICAL TRIAL: NCT06179368
Title: Thyoid Dysfucntion; Does it Affect the Short Term Outcome of Heptic Failure Patiens ?
Brief Title: Throid Dysfunction in Liver Failure and Its Eddects Upon Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, professor, Assiut University
Other Study IDs: IRB121223
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Encephalopathy; Hepatic Impairment; Hypothyroidism; Hepatic Failure
Keywords: Hepatic Failure; Hypothyroidism
MeSH Terms: conditions — Hepatic Encephalopathy; Hypothyroidism; Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothroid group: throid fuction will be evaluated on admission of hepatic failure patients, and the hypothroid patients will be enroled in this group.
  Interventions: Diagnostic Test: hypothroidism
- Euthroid group: throid fuction will be evaluated on admission of hepatic failure patients, and the euothroid patients will be enroled in this group.
  Interventions: Diagnostic Test: euothyroid

INTERVENTIONS:
Diagnostic Test: hypothroidism — throid fuction will be evaluated on admission of hepatic failure patients, and the hypothyroid patients will be enroled in this group.
  Groups: Hypothroid group
Diagnostic Test: euothyroid — throid fuction will be evaluated on admission of hepatic failure patients, and the euothyroid patients will be enroled in this group.
  Groups: Euthroid group

SUMMARY:
Liver plays an important role in the metabolism of thyroid hormones, as it is the most important organ in the peripheral conversion of tetraiodothyronine (T4) to triiodothyronine (T3) by Type 1 deiodinase.

DETAILED DESCRIPTION:
In clinical terms, cirrhosis is described as are either "compensated" or "decompensated." Decompensation means cirrhosis complicated by one or more of the following features: jaundice, ascites, hepatic encephalopathy (HE), or bleeding varices. Ascites is the usual first sign. Hepatorenal syndrome, hyponatremia, and spontaneous bacterial peritonitis are also features of decompensation, but in these patients, ascites invariably occurs first. Compensated cirrhotic patients have none of these features.

The liver plays an important role in the metabolism of thyroid hormones, as it is the most important organ in the peripheral conversion of tetraiodothyronine (T4) to T3 by Type 1 deiodinase.

T4 and T3 regulate the basal metabolic rate of all cells, including hepatocytes, and thereby modulate hepatic function. The liver metabolizes the THS and regulates their systemic endocrine effects. Thyroid diseases may perturb liver function; liver disease modulates thyroid hormone metabolism; and a variety of systemic diseases affect both the organs.

ELIGIBILITY:
Inclusion Criteria:

- hepatic fauiure patients

Exclusion Criteria:

* hypethyroid patients

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: all hepatic failutre patients who will be admitted to ICU will be enrolled, and throid function will be assessed. Groupingwil be done based upon throid function
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
short termoutcome | (0 to 30 days)
  mortality during hospitalstay

SECONDARY OUTCOMES:
complications | (0 to 30 days)
  suchas renal affection, bleeding tendency ...etc

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Punekar P, Sharma AK, Jain A. A Study of Thyroid Dysfunction in Cirrhosis of Liver and Correlation with Severity of Liver Disease. Indian J Endocrinol Metab. 2018 Sep-Oct;22(5):645-650. doi: 10.4103/ijem.IJEM_25_18. PMID 30294575
- [Background] McCormick PA. Sherlock's Diseases of the Liver and Biliary System Textbook. Hepatic Cirrhosis. In: Dooley JS, Lok AS, Burroughs AK, Heathcote EJ, editors. 12th ed. Ch. 7. UK: Wiley-Blackwell, A John Wiley and Sons, Ltd; 2011. pp. 103-8.